CLINICAL TRIAL: NCT02938780
Title: Using Behavioral Economics to Achieve Improved Healthy Behavior Outcomes in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: L15-178
Record Dates: First submitted 2016-09-19; First posted 2016-10-19 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer Female
Keywords: Behavioral economics; Breast cancer survivors; nutrition; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The subjects in the control group will receive placebo text messages which will be timed as the intervention group that are unrelated to the study or topics of exercise and nutrition.
  Interventions: Other: placebo text message
- Intervention (Experimental): The subjects in the intervention group will receive text messages with nutrition and physical activity-related information throughout the study period on a daily basis, varying text message.
  Interventions: Other: nutrition physical activity text message

INTERVENTIONS:
Other: placebo text message — The subjects in the control group will receive placebo text messages which will be timed as the intervention group that are unrelated to the study or topics of exercise and nutrition.
  Arms: Control
Other: nutrition physical activity text message — The subjects in the intervention group will receive text messages with nutrition and physical activity-related information throughout the study period on a daily basis, varying text message arrival over a 10 am to 7 pm time frame. The American Cancer Society recommends a set of exercise and nutrition behaviors for cancer survivors based upon developed expert evidence. These behaviors have been structured to achieve healthier lifestyles, improve quality of life and reduced mortality. The intervention will provide via text messaging exemplars and social norms designed to improve compliance with this advice.
  Arms: Intervention

SUMMARY:
Preventing or reducing obesity is one factor that has been hailed as a way to improve quality of life, reduce recurrence, and increase survival rates among breast cancer survivors. An experienced team of multi-disciplinary researchers has developed an innovative and unique approach to encourage enhanced nutrition and exercise behaviors in this population using principles of behavioral economics. In particular, the use of social norms or exemplars has been shown in other applications to be effective, and if successful in this population could be inexpensively scaled up for widespread adoption. The proposed pilot study develops a system of text messages for social/mobile media that will provide ongoing reinforcement of desired behavior in breast cancer survivors. These messages would focus on achieving compliance with the expert-developed nutrition and exercise recommendations of the American Cancer Society. In the main study, 310 breast cancer survivors will be randomly placed in intervention and control groups for the 12 week study. Behavior change will be measured using established measures of self-reported behavior. In a sub-study, 60 of the breast cancer survivor participants will also provide blood and urine samples so changes in biomarkers can be assessed. The impact of the study will be measured by biomarkers and self-reported survey responses.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age: 20-75 years old
* No current pregnancy or lactation
* Was diagnosed with Stage 0-IIIB disease and completed all local and systemic therapy (including Herceptin) at least 3 months prior to entry. Women can be on or off anti-hormone therapy.
* Ambulatory
* Willing to be randomized

Exclusion Criteria:

* Current participation in other treatment (chemo/radiotherapy) clinical trials
* Instructed by doctor not to exercise
* Cannot read English
* Not able to receive text messages

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Urinary levels of 8-OHdG | 3 months
  To measure oxidative stress DNA damage. ug/mmol creatinine

SECONDARY OUTCOMES:
physical activity | 3 months
  Use physical activity survey
Intake of fruit and vegetable behavior | 3 months
  Use food intake record
Self-efficacy | 3 months
  Use Self-efficacy survey
Serum total antioxidant capacity | 3 months
  To measure total antioxidant concentration (mM)

CONTACTS AND LOCATIONS:
Overall Officials: Conrad Lyford, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No